CLINICAL TRIAL: NCT05035251
Title: Glymphatic Pathway in Brain Imaging: Evaluation of MRI Findings
Brief Title: Glymphatic Pathway in Brain Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Dr. Panagiota Manava, Senior physician, Institute of Radiology and Nuclear Medicine, Klinikum Nuernberg, Paracelsus Medical University
Other Study IDs: GP_2021_KNN
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Glymphatic System
Keywords: glymphatic system; imaging of blood brain barrier

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental: patients with a condition
- control: patients without condition

SUMMARY:
To investigate the pathways of Gadolinium-based contrast agent (GBCA) in different brain compartments and evaluate correlations of GBCA enhancement with specific diseases.

DETAILED DESCRIPTION:
To investigate the contrast enhancement in different brain compartments. Until recently, it had been assumed that Gadolinium-based contrast agents do not cross the blood-brain barrier, but delayed imaging revealed signal increase in a number of compartments in the CSF (the perilymph of the inner ear, the internal auditory canal, the Meckel's cave, the suprasellar cistern, the ambient cistern and anterior eye compartment). These findings suggested, that Gadolinium-based contrast agents (GBCA) penetrate into the CSF through the choroid plexus and the aqueous chamber of the eye. MRI has provided the evidence of presence of meningeal lymphatic vessels in human and non-human primates for central nervous system waste clearance. It has been demonstrated that heavily T2-weighted fluid-attenuated inversion recovery (hT2w-FLAIR) MRI detects even very low concentrations of GBCA in the CSF.

The aim of our study is to find specific enhancement patterns in various cerebral compartments in correlation with specific diseases and procedures such as radiation, surgery and drug application in delayed gadolinium imaging. Only patients with a clinical indication for GBCA will be included in this prospective study. Before enrollment, each patient will have provided written informed consent of participation and publication prior to inclusion to the observational study. The scan will be performed as baseline before intravenous contrast administration of a single dose of gadoteric acid 20 minutes and 120 minutes after contrast administration. Whole-brain image stacks will be analyzed on patient basis. Regions of interest for signal intensity measurements will be drawn in various cerebral fluid spaces, the size of the region of interest will depend on the target structure. The following structures should be measured: lateral and central aqueous chamber and vitreous body of the eye, distal optic nerve sheath, Meckel's cave, lateral ventricles and basal cisterns.

Data will be expressed as mean values +/- one-fold standard deviation (SD). The normality of data distribution will be assessed using Levene's test. Data showing a Gaussian distribution will be evaluated by an analysis of variances (ANOVA) with a post-hoc analysis. Estimated sample size is around 30 patients in the control and the experimental group. Cases with missing or unavailable data will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with a clinical indication for GBCA
* Written informed consent
* No allergies to GBCA

Exclusion Criteria:

* Contraindications for MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients of a primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-11-11 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of Signal-Intensity (SI)-Measurements with ROI in 3 specific MRI Scans | Baseline (nativ scan), 20 minutes and 120 minutes after contrast media application
  Regions of interest for signal intensity measurements will be drawn in various cerebral fluid spaces, the size of the region of interest will depend on the target structure. Following structures will be measured: lateral and central aqueous chamber and vitreous body of the eye, distal optic nerve sheath, Meckel's cave, lateral ventricles and basal cisterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Radiology and Nuclear Medicine, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deike-Hofmann K, Reuter J, Haase R, Paech D, Gnirs R, Bickelhaupt S, Forsting M, Heussel CP, Schlemmer HP, Radbruch A. Glymphatic Pathway of Gadolinium-Based Contrast Agents Through the Brain: Overlooked and Misinterpreted. Invest Radiol. 2019 Apr;54(4):229-237. doi: 10.1097/RLI.0000000000000533. PMID 30480554
- [Background] Taoka T, Naganawa S. Gadolinium-based Contrast Media, Cerebrospinal Fluid and the Glymphatic System: Possible Mechanisms for the Deposition of Gadolinium in the Brain. Magn Reson Med Sci. 2018 Apr 10;17(2):111-119. doi: 10.2463/mrms.rev.2017-0116. Epub 2018 Jan 25. PMID 29367513
- [Background] Absinta M, Ha SK, Nair G, Sati P, Luciano NJ, Palisoc M, Louveau A, Zaghloul KA, Pittaluga S, Kipnis J, Reich DS. Human and nonhuman primate meninges harbor lymphatic vessels that can be visualized noninvasively by MRI. Elife. 2017 Oct 3;6:e29738. doi: 10.7554/eLife.29738. PMID 28971799
- [Background] Rennels ML, Gregory TF, Blaumanis OR, Fujimoto K, Grady PA. Evidence for a 'paravascular' fluid circulation in the mammalian central nervous system, provided by the rapid distribution of tracer protein throughout the brain from the subarachnoid space. Brain Res. 1985 Feb 4;326(1):47-63. doi: 10.1016/0006-8993(85)91383-6. PMID 3971148
- [Background] Iliff JJ, Wang M, Liao Y, Plogg BA, Peng W, Gundersen GA, Benveniste H, Vates GE, Deane R, Goldman SA, Nagelhus EA, Nedergaard M. A paravascular pathway facilitates CSF flow through the brain parenchyma and the clearance of interstitial solutes, including amyloid beta. Sci Transl Med. 2012 Aug 15;4(147):147ra111. doi: 10.1126/scitranslmed.3003748. PMID 22896675
- [Background] Bedussi B, Almasian M, de Vos J, VanBavel E, Bakker EN. Paravascular spaces at the brain surface: Low resistance pathways for cerebrospinal fluid flow. J Cereb Blood Flow Metab. 2018 Apr;38(4):719-726. doi: 10.1177/0271678X17737984. Epub 2017 Oct 17. PMID 29039724
- [Background] Smith AJ, Yao X, Dix JA, Jin BJ, Verkman AS. Test of the 'glymphatic' hypothesis demonstrates diffusive and aquaporin-4-independent solute transport in rodent brain parenchyma. Elife. 2017 Aug 21;6:e27679. doi: 10.7554/eLife.27679. PMID 28826498
- [Background] Dobson H, Sharp MM, Cumpsty R, Criswell TP, Wellman T, Finucane C, Sullivan JM, Weller RO, Verma A, Carare RO. The perivascular pathways for influx of cerebrospinal fluid are most efficient in the midbrain. Clin Sci (Lond). 2017 Nov 13;131(22):2745-2752. doi: 10.1042/CS20171265. Print 2017 Nov 15. PMID 29021222
- [Background] Iliff JJ, Wang M, Zeppenfeld DM, Venkataraman A, Plog BA, Liao Y, Deane R, Nedergaard M. Cerebral arterial pulsation drives paravascular CSF-interstitial fluid exchange in the murine brain. J Neurosci. 2013 Nov 13;33(46):18190-9. doi: 10.1523/JNEUROSCI.1592-13.2013. PMID 24227727
- [Derived] Manava P, Eckrich C, Luciani F, Schmidbauer J, Lell MM, Detmar K. Glymphatic System in Ocular Diseases: Evaluation of MRI Findings. AJNR Am J Neuroradiol. 2022 Jul;43(7):1012-1017. doi: 10.3174/ajnr.A7552. Epub 2022 Jun 30. PMID 35772805